CLINICAL TRIAL: NCT05887453
Title: An Exploratory Clinical Study to Evaluate the Specificity of Magnetocardiogram in Atrial Fibrillation and the Prediction of Recurrence
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: JWang
Record Dates: First submitted 2023-03-26; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Magnetocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Persistent AF
  Interventions: Device: Magnetocardiography
- Group 2 : Paroxysmal AF
  Interventions: Device: Magnetocardiography
- Healthy controls
  Interventions: Device: Magnetocardiography

INTERVENTIONS:
Device: Magnetocardiography — Magnetocardiography is a device used to exam the dynamic magnetic map of the heart for the diagnosis of some heart diseases

SUMMARY:
This is a prospective, observational clinical study with150 patients of persistent AF (trial group 1), 150 patients of paroxysmal AF (trial group 2), and 150 healthy subjects (control group). The trial is divided into two parts. The aim of first part is to evaluate the sensitivity and specificity of magnetocardiography on diagnosing persistent AF, and the second part is to evaluate the independent predictors of magnetocardiography on predicting recurrence of paroxysmal AF. The patients who had been diagnosed with AF in OPD or IPD will be included. After signing the informed consent letter, medical history of all subjects will be collected, including magnetic cardiogram, 12-lead electrocardiogram, holter electrocardiogram, cardiac ultrasound and blood tests. Patients with paroxysmal AF will be followed up for 3 months, and the recurrence of AF is the observation end point.

ELIGIBILITY:
Group: Group 1 (Persistent AF)

Inclusion criteria：

* Persistent AF is recorded by ECG before the examination of the magnetocardiogram;
* Detailed clinical records, including medical history, cardiovascular risk factors, blood tests, and antiarrhythmic drug therapy;
* It is recommended that antiarrhythmic drugs be discontinued at least 5 days before the examination and continue if atrial fibrillation occurs or the symptoms of atrial fibrillation are obvious;

Exclusion criteria:

* Severe valvular heart disease, structural heart disease, heart function classification ≥ New York Heart Association functional class II, history of ischemic heart disease, left ventricular ejection fraction < 50%, hyperthyroidism, primary pulmonary hypertension, and respiratory disease;
* Patients after radiofrequency ablation;
* The implanted devices in the body effect the magnetic signal during the detection process, such as prosthetic limbs, heart stents or valves contain metal material.
* Unable to maintain the supine position during the examination.

Group: Group 2 (Paroxysmal AF)

Inclusion criteria:

* Persistent AF is recorded by ECG before the examination of the magnetocardiogram;
* Detailed clinical records, including medical history, cardiovascular risk factors, blood tests, and antiarrhythmic drug therapy;
* It is recommended that antiarrhythmic drugs be discontinued at least 5 days before the examination and continue if atrial fibrillation occurs or the symptoms of atrial fibrillation are obvious;

Exclusion criteria:

* Severe valvular heart disease, structural heart disease, heart function classification ≥ New York Heart Association functional class II, history of ischemic heart disease, left ventricular ejection fraction < 50%, hyperthyroidism, primary pulmonary hypertension, and respiratory disease;
* Patients after radiofrequency ablation;
* The implanted devices in the body effect the magnetic signal during the detection process, such as prosthetic limbs, heart stents or valves contain metal material.
* Unable to maintain the supine position during the examination.

Group: Control group

Inclusion criteria:

* No history of AFor other arrhythmias;
* Detailed clinical records, including medical history and cardiovascular risk factors;

Exclusion criteria:

* severe valvular heart disease, structural heart disease,heart function classification ≥ New York Heart Association functional class II, history of ischemic heart disease, left ventricular ejection fraction < 50%, hyperthyroidism, primary pulmonary hypertension, and respiratory disease;
* The implanted devices in the body effect the magnetic signal during the detection process, such as prosthetic limbs, heart stents or valves contain metal material.
* Unable to maintain the supine position during the examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with atrial fibrillation and healthy people without arrhythmia
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2023-03-22 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
sensitivity and specificity | 24 hours
  The sensitivity and specificity of magnetocardiography in the diagnosis of persistent AF
Independent predictors of recurrence of paroxysmal atrial fibrillation | 3 months
  A statistical model is used to obtain the magnetocardiographic parameters that could predict the recurrence of paroxysmal atrial fibrillation.

CONTACTS AND LOCATIONS:
Overall Officials: Jian'an Wang, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No